CLINICAL TRIAL: NCT07174466
Title: Enhanced Digital Access to Bridge Social Needs and Reduce Health Disparities: The e-SINCERE Study
Brief Title: The e-SINCERE Study
Acronym: e-SINCERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Wallace (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Andrea Wallace, Professor, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00181891; 1R01NR021501-01 (NIH)
Record Dates: First submitted 2025-09-12; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Social Determinants of Health (SDOH); Digital Health Literacy; Health Services Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Masking Description: Services to which participants are referred will not be aware of the participant's inclusion in the research study or their study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Control - Standard Referral to 211 (Active Comparator): Participants receive usual care plus a referral to United Way 211 for assistance with social needs. No additional study-provided phone or navigation support is given.
  Interventions: Other: Standard Referral to 211
- Arm 2: Phone - Bridge Phone to 211 (Experimental): Participants receive a study-provided cellphone to ensure stable phone access. They are connected by phone to United Way 211 for assistance with social needs.
  Interventions: Behavioral: e-SINCERE (Phone Support)
- Arm 3: Navigation - Digital Navigator + 211 (Experimental): Participants receive a study-provided cellphone and direct support from a Digital Navigator. The Navigator assists participants in accessing United Way 211 and helps troubleshoot barriers to connecting with services.
  Interventions: Behavioral: e-SINCERE (Digital Navigation)

INTERVENTIONS:
Other: Standard Referral to 211 — Participants receive a standard referral to United Way 211 for assistance with social needs. 211 specialists contact referred patients, provide available service referrals, and follow up in an ad-hoc manner as per standard 211 protocols.
  Arms: Arm 1: Control - Standard Referral to 211
Behavioral: e-SINCERE (Phone Support) — Participants receive a study-provided cellphone to ensure stable phone access. Using this device, participants are connected to United Way 211 specialists, who provide referral services for identified social needs. This intervention focuses on overcoming communication barriers that might otherwise prevent successful service connection.
  Arms: Arm 2: Phone - Bridge Phone to 211
Behavioral: e-SINCERE (Digital Navigation) — Participants receive a study-provided TracFone and direct support from a trained Digital Navigator. The Digital Navigator assists participants with accessing United Way 211 services, troubleshooting barriers to phone or internet use, and reinforcing follow-through on referrals. This arm is designed to provide enhanced, structured navigation support to address digital access barriers and increase successful service connections.
  Arms: Arm 3: Navigation - Digital Navigator + 211

SUMMARY:
The e-SINCERE study will evaluate whether providing stable cell phones and digital navigation assistance helps patients overcome ICT barriers and connect more successfully with community services. The study will begin with patients in the UHealth ED, with additional sites added in the future, and will involve working with community service providers and policy leaders to refine and implement the intervention. Findings from this study may guide the development of future programs and policies to improve access to services for patients facing economic and technological barriers.

ELIGIBILITY:
Inclusion Criteria:

* Community Advisory Board Members

Health system, governmental, and community service stakeholders

Able to understand English

Adult (> 18 years)

- General screening population:

Any patient who completes the SINCERE screener.

Able to understand or read English or Spanish.

- Survey study inclusion criteria:

Any patient who completes the SINCERE screener who has connected with 211 for service outreach

Able to understand or read English or Spanish.

Adult (> 18 years)

Exclusion Criteria:

* Those unable to communicate verbally in English or Spanish
* Those living in nursing facilities, or those who are not otherwise responsible for self-care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Successful connection to community social services (any service) | 6 months after randomization
  Proportion of participants who have at least one documented successful connection to a community social service (e.g., housing assistance, utilities, food support, transportation) within 6 months. Successful connection is defined as a recorded positive outcome in 211 or ServicePoint (client reached and service initiated) or participant self-report confirmed by case notes.

SECONDARY OUTCOMES:
Health-related quality of life (PROMIS Global Health) | Baseline, 2 weeks, 3 months, and 6 months after randomization
  Change in PROMIS Global Health T-score from baseline to 6 months. Higher scores indicate better overall physical and mental health. Analysis will compare mean change between arms.
Emergency department utilization (all-cause ED visits) | 6 months after randomization
  Number of all-cause ED visits per participant during the 6-month follow-up period, obtained from the institution's EDW and participant self-report for non-UHealth visits. Analysis will compare mean visits and proportion with any ED revisit between arms.
Digital access stability (phone connectivity) | 6 months after randomization
  Proportion of participants in the phone/navigation arms with continuous phone connectivity (TracFone active and reachable) for at least 5 of 6 months. Connectivity assessed via phone service logs and navigator contact attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wallace, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No